CLINICAL TRIAL: NCT00797641
Title: European Survey of Non-Variceal Upper Gastro Intestinal Bleeding
Brief Title: European Survey of Non-Variceal Upper Gastro Intestinal Bleeding (NVUGIB)
Acronym: ENERGIB
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Dr Rick Lones, BM MRCGP MFPM DRCOG DFFP, European Medical Affairs Director, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-GEU-DUM-2008/2
Record Dates: First submitted 2008-11-21; First posted 2008-11-25 (Estimated); Last update posted 2009-12-04 (Estimated); Status verified 2009-12

CONDITIONS: Non-variceal Upper Gastrointestinal Bleeding; Gastrointestinal Ulcer; Gastrointestinal Hemorrhage
Keywords: bleeding; ulcer; hemorrhage; gastrointestinal diseases; digestive system disease; peptic ulcer; proton pump inhibitor
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Hemorrhage; Ulcer; Gastrointestinal Diseases; Digestive System Diseases; Peptic Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients admitted to the hospital, or inpatients admitted for another reason, presenting with overt non-variceal upper GI bleed manifesting as hematemesis/coffee ground vomiting, melena, hematochezia, as well as other clinical or laboratory evidence of acute blood loss from the upper gastrointestinal tract

SUMMARY:
The aim of this study is to assess the current management strategies in a pan-European "real-life" setting to uncover the unmet need in this area: non-variceal gastrointestinal bleedings.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the hospital or inpatients with an overt non-variceal upper GI bleed manifesting as hematemesis/coffee ground vomiting, melena, hematochezia, as well as other clinical/laboratory evidences of acute blood loss from the upper GI tract
* Evidence that an upper GI endoscopy was performed
* The complete medical record is available for study related hospitalization.

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the hospital, or inpatients admitted for another reason, presenting with overt non-variceal upper GI bleed manifesting as hematemesis/coffee ground vomiting, melena, hematochezia, as well as other clinical or laboratory evidence of acute blood loss from the upper gastrointestinal tract
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To describe clinical outcomes associated with current strategies of endoscopic and pharmacological treatment in several European countries, in respect of bleeding continuation, rebleeding, surgery and in-hospital mortality | Up to 30 days after the episode (bleeding)

SECONDARY OUTCOMES:
To describe clinical management and how this compares across countries and Hospital types | Up to 30 days after the episode (bleeding)
To assess predictive factors for clinical management strategies and predictive factors related to clinical outcomes | Up to 30 days after the episode (bleeding)
To assess health care resource consumption in patients admitted with non-variceal upper gastrointestinal bleeding and the main drivers | Up to 30 days after the episode (bleeding)

CONTACTS AND LOCATIONS:
Overall Officials: Ángel Lanas, MD, Principal Investigator — Hospital Clínico Universitario Lozano Blesa, Zaragoza (Spain); Javier N Rivero, MSc, Study Director — Medical Department, AstraZeneca Spain
Locations (97):
- Belgium (25):
  - Research site, Aalst
  - Research site, Anderlecht
  - Research site, Assebroek
  - Research site, Braine-l'Alleud
  - Research site, Brasschaat
  - Research site, Bruges
  - Research site, Brussels
  - Research site, Charleroi
  - Research site, Deurne
  - Research site, Edegem
  - Research site, Geraardsbergen
  - Research site, Ghent
  - Research site, Hasselt
  - Research site, Herentals
  - Research site, Kortrijk
  - Research site, Lier
  - Research site, Liège
  - Research site, Mechelen
  - Research site, Ottignies Lln
  - Research site, Tielt
  - Research site, Tournai
  - Research site, Turnhout
  - Research site, Wetteren
  - Research site, Wilrijk
  - Research site, Zottegem
- Greece (3):
  - Research site, Athens
  - Research site, Larissa
  - Research site, Thessaloniki
- Italy (12):
  - Research site, Bolzano
  - Research site, Cosenza
  - Research site, Crema
  - Research site, Forlì
  - Research site, Milan
  - Research site, Napoli
  - Research site, Novara
  - Research site, Revenna
  - Research site, Roma
  - Research site, S. Giovanni Rotondo
  - Research site, Siena
  - Research site, Trieste
- Norway (14):
  - Research site, Arendel
  - Research site, Ålesund
  - Research site, Bodø
  - Research site, Drammen
  - Research site, Fredrikstad
  - Research site, Kristiansand
  - Research site, Levanger
  - Research site, Lillehammer
  - Research site, Oslo
  - Research site, Rud
  - Research site, Stavanger
  - Research site, Tromsø
  - Research site, Trondheim
  - Research site, Tønsberg
- Portugal (11):
  - Research site, Almada
  - Research site, Angra do Heroísmo
  - Research site, Braga
  - Research site, Caldas da Rainha
  - Research site, Castelo Branco
  - Research site, Covilha
  - Research site, Funchal
  - Research site, Leiria
  - Research site, Ponta Delgada
  - Research site, Santarém
  - Research site, Torres Novas
- Spain (20):
  - Research site, Alcázar de San Juan
  - Research site, Alicante
  - Research site, Barcelona
  - Research site, Burgos
  - Research site, Córdoba
  - Research site, Huesca
  - Research site, La Cuesta de Arguijon
  - Research site, Las Palmas de Gran Canaria
  - Research site, Logroño
  - Research site, Madrid
  - Research site, Marbella
  - Research site, Murcia
  - Research site, Ourense
  - Research site, Oviedo
  - Research site, Pamplona
  - Research site, Sabadell
  - Research site, Santiago de Compostela
  - Research site, Seville
  - Research site, Valencia
  - Research site, Zaragoza
- Turkey (Türkiye) (12):
  - Research site, Ankara
  - Research site, Antalya
  - Research site, Batman
  - Research site, Bursa
  - Research site, Diyarbakır
  - Research site, Elâzığ
  - Research site, Gaziantep
  - Research site, Istanbul
  - Research site, Izmir
  - Research site, Konya
  - Research site, Malatya
  - Research site, Mersin

REFERENCES:
- [Derived] Lanas A, Aabakken L, Fonseca J, Mungan Z, Papatheodoridis G, Piessevaux H, Rotondano G, Nuevo J, Tafalla M. Variability in the management of nonvariceal upper gastrointestinal bleeding in Europe: an observational study. Adv Ther. 2012 Dec;29(12):1026-36. doi: 10.1007/s12325-012-0069-x. Epub 2012 Dec 6. PMID 23225523
- [Derived] Mungan Z. An observational European study on clinical outcomes associated with current management strategies for non-variceal upper gastrointestinal bleeding (ENERGIB-Turkey). Turk J Gastroenterol. 2012;23(5):463-77. doi: 10.4318/tjg.2012.0402. PMID 23161291
- [Derived] Lanas A, Aabakken L, Fonseca J, Mungan ZA, Papatheodoridis GV, Piessevaux H, Cipolletta L, Nuevo J, Tafalla M. Clinical predictors of poor outcomes among patients with nonvariceal upper gastrointestinal bleeding in Europe. Aliment Pharmacol Ther. 2011 Jun;33(11):1225-33. doi: 10.1111/j.1365-2036.2011.04651.x. Epub 2011 Apr 11. PMID 21480935